CLINICAL TRIAL: NCT01167296
Title: Safety of Leaving Cook Balloon Uterine Stent in Uterus for One Month
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shin Kong Wu Ho-Su Memorial Hospital (Other)
Responsible Party: Principal Investigator, Yu-Hung Lin, MD, Shin Kong Wu Ho-Su Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SKH-8302-99-DR-27
Record Dates: First submitted 2010-07-21; First posted 2010-07-22 (Estimated); Last update posted 2013-06-10 (Estimated); Status verified 2013-06

CONDITIONS: Intrauterine Adhesion
Keywords: Intrauterine adhesion; Cook balloon uterine stent
MeSH Terms: conditions — Gynatresia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cook balloon uterine stent (Active Comparator): Immediately before hysteroscopic surgery, a culture tip is inserted into the uterine cavity and sent for culture. Another culture was done 30 days later, and a second-look hysteroscope is done to evaluate the healing of uterine cavity.removed uterine stent was sent for bacterial culture too.
  Interventions: Device: Cook balloon uterine stent
- without Cook balloon uterine stent (Experimental): Immediately before hysteroscopic surgery, a culture tip is inserted into the uterine cavity and sent for culture. Another culture was done 30 days later, and a second-look hysteroscope is done to evaluate the healing of uterine cavity.
  Interventions: Device: Cook balloon uterine stent

INTERVENTIONS:
Device: Cook balloon uterine stent — Immediately before hysteroscopic surgery, a culture tip is inserted into the uterine cavity and sent for culture. Another culture was done 30 days later, and a second-look hysteroscope is done to evaluate the healing of uterine cavity.

SUMMARY:
To use Cook balloon uterine stent to prevent intrauterine adhesion (IUA), and to see if leaving it in the uterus will cause uterine infection.

DETAILED DESCRIPTION:
Background：Intrauterine adhesion (IUA) can cause infertility. Hysteroscopic surgery can effectively treat most IUA. In order to prevent adhesion reformation after surgery, most gynecologists will prescribe high-dose estrogen to stimulate endometrial growth, and leave an IUD or a Foley catheter in uterus for 1-3 months. But neither IUD nor Foley catheter conform to the uterine cavity. The Cook balloon uterine stent was designed to fit into the uterine cavity. But it was designed to tamponade the uterus to prevent post-operative uterine bleeding. It's not known if it can be left in the uterus for 30 days.

Study Design：Uterine culture was done before hysteroscopic surgery, and 30 days later. The study group comprise patients with uterine stent; the control group comprise patients who undergo hysteroscopic surgeries but without uterine stent.

Method：Immediately before hysteroscopic surgery, a culture tip is inserted into the uterine cavity and sent for culture. Another culture was done 30 days later, and a second-look hysteroscope is done to evaluate the healing of uterine cavity. The removed uterine stent was sent for bacterial culture too. The same procedures are done for patients with and without uterine stent. The bacterial counts will be compared before and after hysterosocpic surgeries, and between the two groups of patients.

Effect：If leaving the uterine stent in the uterus up to 30 days does not cause bacteria to grow, we can be confident to leave the stent for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* intrauterine adhesion women

Exclusion Criteria:

* allergic to Cook balloon uterine stent

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-07; Primary Completion 2011-07 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
intrauterine bacteria count | one year

SECONDARY OUTCOMES:
intrauterine adhesion | one year

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Obstetrics and Gynecology, Shin-Kong Wu-Ho-Su Memerial Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Lin YH, Jang TN, Hwang JL, Huang LW, Seow KM, Hsieh BC, Huang CH. Bacterial colonization with balloon uterine stent placement in the uterus for 30 days: a randomized controlled clinical trial. Fertil Steril. 2015 Feb;103(2):513-8.e2. doi: 10.1016/j.fertnstert.2014.10.032. Epub 2014 Nov 20. PMID 25467040